## EH21-338: Observational and Prospective Study on the Performance of Inherited Risk Assessment for Predicting Prostate Cancer from Prostate Biopsy (GenBx)

PI: Jianfeng Xu, MD, DrPH

Version 1

Created: 12/12/2021

Prospective study on the performance of inherited risk assessment for predicting prostate cancer from prostate biopsy

## Analytical plan

Outcome variable: Diagnosis of PCa from prostate biopsy.

Inherited risk assessment: Rare pathogenic mutations (RPMs) in 11 guideline-recommended genes and genetic risk score (GRS) based on published GWAS (genome-wide association studies)-significant SNPs. Patients will be classified into three groups based on inherited risk: high-risk (RPMs+ and/or GRS ≥1.5), low-risk (RPMs- and GRS <1.5), and intermediate-risk (remaining subjects).

**Other variables**: Age, race/ethnicity, body mass index (BMI), PSA, as well as Prostate Health Index and MRI results if they are available.

**Blind design**: Prostate biopsy will be performed prior to inherited risk assessment. Inherited risk assessment will be performed blinded to the biopsy outcomes.

## Data analysis:

- 1. Descriptive analysis of prostate cancer detection rate in three inherited risk groups.
- 2. Trend test for higher prostate cancer detection rate in patients with increasing inherited risk (low, intermediate, and high) using a chi-square test for linear trend.
- 3. Association of inherited risk (high vs. remaining) with diagnosis of prostate cancer using multivariate logistic regression adjusting for age, race, BMI, and PSA.